CLINICAL TRIAL: NCT06415630
Title: Multiple Automated Machine-learning Prediction Models for Postoperative Reintubation in Patients With Acute Aortic Dissection
Brief Title: Prediction Models for Postoperative Reintubation in Patients With Acute Aortic Dissection
Acronym: ADreintubate
Status: Completed | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: WHUH-AADreintu
Record Dates: First submitted 2024-05-09; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Nomogram; Prediction Model; Type A Aortic Dissection; Postoperative Reintubation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- training group: To determine potential predictive factors, the training group was subjected to LASSO regression analysis, which effectively eliminated several irrelevant or multicollinearity independent variables to reduce high-dimensional data.Seven models were initially constructed in the training group: multivariable logistics regression (MLR), decision-tree modeling, random forest, XGBoost, Support Vector Machines, k-nearest neighbors, and LightGBM.
  Interventions: Procedure: Type A aortic dissection surgery
- testing group: Testing group was used to examine the performance of the seven prediction models, including discrimination and calibration performance. Finally, the model with best discrimination and calibration performance was used to construct nomogram for predicting reintubation.
  Interventions: Procedure: Type A aortic dissection surgery

INTERVENTIONS:
Procedure: Type A aortic dissection surgery — Patients with type A aortic dissection undergone surgery.

SUMMARY:
Reintubation is an adverse postoperative complication in patients with Type A aortic dissection (AAD) that correlates to poor outcomes. This study aims to analyze the risk factors associated with reintubation and to create a fully automated score model to predict the incidence of reintubation. A total of 861 patients diagnosed with AAD and undergoing surgical procedures in a single institution between January 2018 and October 2023 were selected in wuhan Union Hospital. Preoperative and postoperative informmation was used for seeking risk factors and build prediction model for postoperative reintubation. Finally, 5 risk factors wasidentified and a nomogram was established for predicting postoperative reintubation in patients with AAD.

ELIGIBILITY:
Inclusion Criteria:

(1) patients diagnosed with AAD admitted for open surgery; (2) aged 18 years or older.

Exclusion Criteria:

(1) patients deceased during or within 24 hours after surgery; (2) patients with preoperative intubation.

Ages: 19 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A total of 892 patients with AAD who underwent open surgery at Wuhan Union Hospital between January 2018 and October 2023 were enrolled using a convenient sampling method.
Sampling Method: Probability Sample
Enrollment: 861 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
postoperative reintubation | 3 month
  reintubation incidence in patients with type A aortic dissection undergoing surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No